CLINICAL TRIAL: NCT02394964
Title: The Human Microbiome in Immune-Mediated Diseases
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Arthritis Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1408014402; U01AI101990 (NIH); R01AI118855-01 (NIH)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Autoimmune
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, oral swab, skin swab, stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Systemic Lupus Erythematosus: Blood, stool, and swab samples will be collected at baseline, week 4, and week 8 and compared with control samples
  Interventions: Other: Sample Collection
- Subacute Cutaneous Lupus Erythematosus: Blood, stool, and swab samples will be collected at baseline, week 4, and week 8 and compared with control samples
  Interventions: Other: Sample Collection
- Control: Blood, stool, and swab samples will be collected for comparison to each disease group
  Interventions: Other: Sample Collection
- Cutaneous T-Cell Lymphoma: Blood and swab samples will be collected for comparison to each disease group
  Interventions: Other: Sample Collection
- Autoimmune Disorders: Blood, stool, and swab samples will be collected for comparison to each disease group
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — Sample collection of blood, stool, and buccal and skin swab samples will be collected at baseline, week 4, and week 8

SUMMARY:
The immune system is influenced by the commensal microbes that live in the gut and on the skin. This study aims to characterize the microbiota of subjects with autoimmune disease in order to determine whether certain microbial species may cause or worsen immune-mediated diseases

DETAILED DESCRIPTION:
This is a combination of a defined pilot microbiome study as well as exploratory mechanistic research with candidate commensals identified based on known structures accessible in public databases. In the observational prospective two-center study, subjects will be followed for 8 weeks. The study will consist of a total of 3 study visits (0, 4 and 8 weeks). Screening and baseline visits (week 0) will take place at the same time. A study window period of +/- 7 days will be allowed for follow-up study visits. The mechanistic in vitro research with subjects' blood cells and candidate commensals will typically require between 2-4 visits for sampling, but will not be limited by the frequency of visits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Diagnosis of an immune-mediated disease by a healthcare provider, including but not limited to: systemic lupus erythematosus, subacute cutaneous lupus erythematosus

Exclusion criteria for pilot study (subjects enrolled in the exploratory mechanistic study arm will not be required to meet exclusion criteria and may be enrolled if the investigators believe that the subject can help address the scientific aim)..

Exclusion Criteria:

* Ongoing chronic infection (viral, bacterial or fungal) including known HIV, Hepatitis B/C
* Acute infection receiving any antibiotics or any use of antibiotics within 90 days prior to screening
* For skin swab collection (see also appendix D):

  * No use of topical antibiotics within 7-days prior to collection of swab, other than use in normal hand washing.
  * No use of topical antimicrobial products (as outlined in appendix F) within 48 hours prior to collection of swab
  * Subject must not have bathed within 8-hours of swab collection.
* For oral swab collection (see also appendix D):

  * No use of antiseptic mouth washes (as outlined in appendix F) within 48 hours of swab collection
  * Subjects must not have brushed teeth or flossed within 8-hours of swab collection
* Major gastrointestinal surgery less than 5 years prior to enrollment (with the exception of appendectomy)
* Any Gastrointestinal bleeding history
* Inflammatory Bowel Disease diagnosed by biopsy
* Bulimia or anorexia nervosa
* Probiotics (greater than estimated 109 cfu or organisms per day) within 90 days prior to enrollment (with the exception of fermented beverages, milks or yogurts).
* Morbid obesity (BMI ≥ 40)
* Type I Diabetes Mellitus
* Diabetes Mellitus type 2, poorly controlled defined as Hgb A1c greater than 8% on medical therapy
* Malignancy within one year prior to screening (with the exception of non-metastatic squamous or basal cell skin carcinomas and cervical carcinoma if received curative surgical treatment)
* Known illicit drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with immune-mediated disorders including but not limited to: systemic lupus, cutaneous lupus, Sjogren's Syndrome, mixed connective tissue disease, dermatomyositis/polymyositis, celiac sprue with or without dermatitis herpetiformis, scleroderma, ANCA-associated vasculitis
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-11; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Difference in Commensal bacteria | 8 weeks
  Difference in disease group vs. control commensal bacteria will be compared by looking at the relative abundances of the microbiota

SECONDARY OUTCOMES:
Immune Cross-reactivity with commensal bacteria | 8 weeks
  T and B cells in patients with immune-mediated diseases will cross react with specific microbial antigens

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kriegel, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruff WE, Greiling TM, Kriegel MA. Host-microbiota interactions in immune-mediated diseases. Nat Rev Microbiol. 2020 Sep;18(9):521-538. doi: 10.1038/s41579-020-0367-2. Epub 2020 May 26. PMID 32457482
- [Result] Zegarra-Ruiz DF, El Beidaq A, Iniguez AJ, Lubrano Di Ricco M, Manfredo Vieira S, Ruff WE, Mubiru D, Fine RL, Sterpka J, Greiling TM, Dehner C, Kriegel MA. A Diet-Sensitive Commensal Lactobacillus Strain Mediates TLR7-Dependent Systemic Autoimmunity. Cell Host Microbe. 2019 Jan 9;25(1):113-127.e6. doi: 10.1016/j.chom.2018.11.009. Epub 2018 Dec 20. PMID 30581114
- [Result] Ruff WE, Dehner C, Kim WJ, Pagovich O, Aguiar CL, Yu AT, Roth AS, Vieira SM, Kriegel C, Adeniyi O, Mulla MJ, Abrahams VM, Kwok WW, Nussinov R, Erkan D, Goodman AL, Kriegel MA. Pathogenic Autoreactive T and B Cells Cross-React with Mimotopes Expressed by a Common Human Gut Commensal to Trigger Autoimmunity. Cell Host Microbe. 2019 Jul 10;26(1):100-113.e8. doi: 10.1016/j.chom.2019.05.003. Epub 2019 Jun 18. PMID 31227334
- [Result] Greiling TM, Dehner C, Chen X, Hughes K, Iniguez AJ, Boccitto M, Ruiz DZ, Renfroe SC, Vieira SM, Ruff WE, Sim S, Kriegel C, Glanternik J, Chen X, Girardi M, Degnan P, Costenbader KH, Goodman AL, Wolin SL, Kriegel MA. Commensal orthologs of the human autoantigen Ro60 as triggers of autoimmunity in lupus. Sci Transl Med. 2018 Mar 28;10(434):eaan2306. doi: 10.1126/scitranslmed.aan2306. PMID 29593104
- [Result] Manfredo Vieira S, Hiltensperger M, Kumar V, Zegarra-Ruiz D, Dehner C, Khan N, Costa FRC, Tiniakou E, Greiling T, Ruff W, Barbieri A, Kriegel C, Mehta SS, Knight JR, Jain D, Goodman AL, Kriegel MA. Translocation of a gut pathobiont drives autoimmunity in mice and humans. Science. 2018 Mar 9;359(6380):1156-1161. doi: 10.1126/science.aar7201. PMID 29590047
- [Derived] Zhou H, Balint D, Shi Q, Vartanian T, Kriegel MA, Brito I. Lupus and inflammatory bowel disease share a common set of microbiome features distinct from other autoimmune disorders. Ann Rheum Dis. 2025 Jan;84(1):93-105. doi: 10.1136/ard-2024-225829. Epub 2025 Jan 2. PMID 39874239